CLINICAL TRIAL: NCT01714583
Title: The Relationship Between Positive End Expiratory Pressure and Cardiac Index in Patients With ARDS Managed on a Fluid Protocol: A Secondary Analysis of a Prospective Trial
Brief Title: The Relationship Between Positive End Expiratory Pressure and Cardiac Index in Patients With Acute Respiratory Distress Syndrome (ARDS) Managed on a Fluid Protocol
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: NHLBI T32 HL007106-34
Record Dates: First submitted 2012-10-19; First posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Mechanical ventilation; ARDS; acute lung injury; cardiac function; cardiac index; heart-lung interaction
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High PEEP: Cohort of participants with positive end-expiratory pressure (PEEP) greater than or equal to 12cm.
- Low PEEP: Cohort of participants with positive end-expiratory pressure (PEEP) less than 12cm.

SUMMARY:
The objective of this study is to evaluate the association between positive end-expiratory pressure (PEEP) setting and cardiac function, as measured by cardiac index, in patients with acute respiratory distress syndrome (ARDS) who were managed on the NHLBI ARDS Network Fluid and Catheter Treatment Trial (FACTT) fluid protocols.

DETAILED DESCRIPTION:
This is a secondary cross-sectional analysis of the FACTT multi-center randomized controlled trial enrolling adult patients within 48 hours of ARDS onset from twenty medical centers across the US, some of which included more than one hospital. We studied the patients who were randomized to the pulmonary artery catheter arm of the FACTT study. The investigators included patients that had PEEP and cardiac index measurements performed within a short period of each other during the first 3 days of the FACTT study enrollment. Since FACTT had a 2x2 factorial design, half of the patients were in a 'liberal fluids' study arm, and the other half were in a 'conservative fluids' study arm.

ELIGIBILITY:
Inclusion Criteria:

Acute lung injury diagnosis (as defined by The American - European Consensus Conference on ARDS) of < 48 hours in duration.

Patients in the Pulmonary Artery catheter (PAC) arm of the FACTT study. PaO2 / FiO2 ratio of < 200. Data from the first 3 days of mechanical ventilation.

Exclusion Criteria:

Select chronic conditions that could independently influence survival (e.g., expected 6-month survival < 50%) and / or ventilator weaning.

PEEP values missing. FiO2 values missing. PaO2 values missing. Cardiac index values missing Pressors and / or inotropes requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a secondary cross-sectional analysis of the FACTT multi-center randomized controlled trial enrolling adult patients within 48 hours of ARDS onset from twenty medical centers across the US, some of which included more than one hospital. We studied the patients who were randomized to the pulmonary artery catheter arm of the FACTT study. We included patients that had PEEP and cardiac index measurements performed within a short period of each other during the first 3 days of the FACTT study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cardiac Index | Cross sectional (i.e. at time Zero only)
  The cardiac index is a cardiodynamic measure based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area to yield the cardiac index.
  The cardiac index which is the outcome measure is assessed at the same time as the PEEP (which is the independent variable) is measured.
  The study participants are NOT followed for any period of time. This is a cross-sectional study design. Both variables (Cardiac index and PEEP) are measured at the same time.

CONTACTS AND LOCATIONS:
Overall Officials: Wassim H Fares, MD MSc, Principal Investigator — Yale University, School of Medicine, Department of Internal Medicine, Section of Pulmonary and Critical Care Medicine
Locations (1):
- Yale University, School of Medicine, Department of Internal Medicine, Section of Pulmonary and Critical Care Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Fares WH, Carson SS; NIH NHLBI ARDS Network. The relationship between positive end-expiratory pressure and cardiac index in patients with acute respiratory distress syndrome. J Crit Care. 2013 Dec;28(6):992-7. doi: 10.1016/j.jcrc.2013.06.021. Epub 2013 Aug 28. PMID 23993772